CLINICAL TRIAL: NCT06256055
Title: A First-In-Human, Single Arm, Open-label, Phase 1 Dose-Escalation Study of UCMYM802 Injection in Mesothelin-positive Advanced Malignant Solid Tumors
Brief Title: Phase 1 Study of UCMYM802 Injection in Mesothelin-positive Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UTC Therapeutics Inc. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCMYM802-Ⅰ
Record Dates: First submitted 2024-01-22; First posted 2024-02-13 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-03

CONDITIONS: Malignant Mesothelioma; Colorectal Cancer; Bile Duct Cancer; Rectal Cancer; Ovary Cancer; Pancreatic Cancer; Breast Cancer Female
Keywords: mRNA CAR-T; Solid tumor; mesothelin
MeSH Terms: conditions — Mesothelioma, Malignant; Colorectal Neoplasms; Bile Duct Neoplasms; Rectal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Accelerated titration design and 3+3 design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCMYM802 Injection (Experimental): Active ingredient：Anti-MSLN CAR+ T cell
  Interventions: Biological: UCMYM802 Injection

INTERVENTIONS:
Biological: UCMYM802 Injection — 1×10^8~2×10^9 cells will be infused intravenously for 4 times.

SUMMARY:
This is a first-in-human, single-arm, open-label, dose escalation clinical study to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic characteristics, immunogenicity and preliminary efficacy of UCMYM802 (Circular mRNA encoding Anti-Mesothelin CAR-T) injection in patients with Mesothelin-positive advanced malignant solid tumors.

DETAILED DESCRIPTION:
All subjects who qualified after screening will receive the proposed dose of UCMYM802 injection once a week, 4 times in total. The Starting Dose of cell injection was set at 1×10^8, and the maximum dose was set at 2.0×10^9.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years old,regardless of gender
2. Diagnosed Patients with malignant solid tumors confirmed histopathologically (including but not limited to mesothelioma, pancreatic cancer, biliary tract cancer, lung cancer, ovarian cancer, gastric cancer, colorectal cancer, thymus cancer, esophageal cancer, breast cancer, and endometrial cancer, etc.) who fail or cannot tolerate standard treatment or lack effective treatment methods as defined by CSCO and NCCN guidelines
3. At least have one evaluable lesion;
4. Patients who Can provide tumor tissue samples or tumor samples can be obtained through methods such as tumor biopsy;
5. Positive expression of MSLN in tumor cells confirmed by Immunohistochemistry (IHC) or immunocytochemistry (ICC) staining
6. Eastern Cooperative Oncology Group (ECOG) performance score at 0 or 1;
7. Life expectancy ≥ 3 months.
8. The organ function must meet the following requirements:

   * Hematological functions: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (Without receiving G-CSF support within 7 days prior to laboratory examination); Absolute Lymphocyte Count (ALC) ≥ 0.5 × 10^9/L; Hemoglobin (HGB) ≥ 80 g/L (without receiving any blood transfusion or erythropoietin stimulating agent therapy within 7 days before the laboratory examination);Platelet count (PLT) ≥ 75 × 10^9/L (Without receiving platelet transfusion and TPO within 7 days before the laboratory examination)；
   * Hepatic functions: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN)(for patients with primary liver tumors or liver metastases ，AST and ALT≤ 5.0× ULN)；Total bilirubin (TBIL) ≤ 1.5 × ULN(for patients with primary liver tumors or liver metastases，TBIL≤ 3.0× ULN；patients with Gilbert's Syndrome，TBIL≤3×ULN and Direct bilirubin≤ 1.5 × ULN).
   * Coagulation functions: Activated partial thromboplastin time (APTT) ≤ 1.5×ULN.
   * Renal functions: Serum creatinine (Cr)≤1.5 × ULN; or Creatinine clearance rate (Ccr) ≥ 60 mL/min（Cockcroft-Gault）.
   * Cardiac functions: Left ventricular ejection fraction (LVEF) > 50% (confirmed by ECHO).
   * Lung fuction:Pulse oxygen saturation (SpO2) > 95% at rest without oxygenation
9. Women of childbearing potential (WCBP) must have negative results on a serum pregnancy test, and WCBP or Male who have partners of reproductive potential must agree to use effective contraceptive methods to avoid pregnancy throughout the screening and study period until 1 year after the last cell infusion;
10. Voluntary signing informed consent form(s) indicating that they are willing to participate in the study and are able to comply with the protocol.

Exclusion Criteria:

1. Have received systemic antitumor therapy involving cytotoxic chemical agents, monoclonal antibodies or immunotherapy within 4 weeks or 5 half-lives (whichever is shorter) prior to signing the informed consent form（ICF）; Have received systemic glucocorticoids (prednisone or other equivalent hormone at a dose ≥ 10 mg/day) or other treatments to suppress the immune system within 2 weeks prior to signing the ICF; Have received systemic antitumor therapy involving biologics or other approved small molecule targeted inhibitors within 1 week or 5 half-lives (whichever is shorter) prior to signing the ICF; Have received treatments with Chinese herbal medicines (CHM) and Chinese proprietary medicines (CPM) that has an antitumor indication within 1 week prior to signing the ICF;
2. Pregnant or lactating women;
3. The finding of Positive hepatitis B surface antigen (HBsAg) or positive hepatitis B core antibody (HBcAb) and the result of quantitative HBV DNA test in peripheral blood is above the lower limit of detection (LLOD); positive Hepatitis C virus (HCV) antibody, and the result of quantitative HCV RNA test in peripheral blood is above the LLOD; The presence of positive Human immunodeficiency virus (HIV) antibody; positive Syphilis antibody test;
4. Patients with Epstein-Barr Virus (EBV) DNA positive.
5. Non-hematologic toxicity due to prior therapy (surgery, chemotherapy, radiation, targeted therapy, and immunotherapy, etc.) have not resolved to ≤ CTCAE grade 1 (except alopecia, peripheral sensory nerve disorders);
6. Have received any prior xenotransplantation of tissues /organs (including bone marrow transplantation, stem cell transplantation, liver transplantation, and kidney transplantation, etc.), except for transplants that do not require immunosuppression (e.g., corneal graft and hair transplantation, etc.);
7. Previoulsly received any anti mesothelin (MSLN) treatment and any genetically modified cell therapy within 6 months prior to signing the informed consent form;
8. Have undergone major surgery and not fully recovered within 4 weeks prior to signing informed consent or have a history of severe trauma that have not recovered, or planned to receive major surgery within 12 weeks after cell infusion;
9. Presence of known CNS metastases
10. Presence of clinically significant systemic disease (e.g., severe active infection or significant dysfunctions of the heart, lungs, liver, nervous system, or other organs) that, at the discretion of the investigator, impairs the patient's ability to tolerate the treatment specified in this trial protocol or significantly increases the risk of complications. Including but not limited to:

    * Presence of uncontrolled severe active infection (e.g., sepsis, bacteremia, and viremia, etc.);
    * Congestive heart failure classified as > class I based on New York Heart Association (NYHA);
    * Clinically significant severe aortic stenosis and symptomatic mitral valve stenosis;
    * QTc > 450 msec or QTc > 480 msec as shown by ECG in patients with bundle branch block;
    * Presence of uncontrolled clinically significant arrhythmias within 6 months prior to signing the ICF;
    * Presence of acute coronary syndrome within 6 months prior to signing the ICF (e.g., unstable angina and myocardial infarction);
    * Hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) or pulmonary hypertension that has not been controlled by medication;
    * Cerebrovascular accident within 6 months prior to signing informed consent, including: Transient ischemic attack (TIA), brain infarction, cerebral hemorrhage and subarachnoid hemorrhage;
    * Presence of active, chronic or relapsing (within 1 year prior to signing the ICF) severe autoimmune disorder or history of immune-mediated disease requiring steroid or other immunosuppressive therapy, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, autoimmune thyroid disorder, and multiple sclerosis, etc. Except: Hypothyroidism that can be controlled by thyroid hormone replacement therapy alone, skin diseases that do not require systemic treatment (e.g. vitiligo and psoriasis), celiac disease that is already under control;
    * Presence of any form of primary or secondary immunodeficiency, such as: Severe combined immunodeficiency (SCID);
    * Possibility of bleeding due to esophageal or gastric varices as judged by the investigator.
11. History of severe systemic hypersensitivity reactions to the drugs/components used in this trial [such as: fludarabine, cyclophosphamide, dimethyl sulfoxide (DMSO), low molecular dextran, and human serum albumin (HSA), etc.];
12. Have received a live attenuated vaccine within 4 weeks prior to signing the ICF;
13. Participation in another clinical trial within 4 weeks prior to signing the ICF(Enrolled and given of investigational drugs/treatments);
14. History of another malignancy within the previous 5 years (except adequately treated non-melanoma skin cancer and in situ cancer in the following sites: breast, stomach, colon, and cervical, etc.);
15. Prior neuropsychiatric disorders diagnosed by International Classification of Diseases 11th Revision (ICD-11) criteria for mental and behavioral disorders or neuropsychiatric disorders to be excluded as assessed by the investigator, including but not limited to epilepsy, schizophrenia, dementia, addictive behaviors due to drugs and alcohol, etc.;
16. Presence of other conditions that, in the judgment of the investigator, would preclude the patient from participating in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Event (TEAE) | 2 years
  Incidence and severity of treatment emergent adverse events.
Treatment Related Adverse Event (TRAE) | 2 years
  Incidence and severity of treatment related adverse events
Adverse Events of Special Interest (AESI) | 2 years
  Incidence and severity of adverse event of special interest
Incidence of Dose-limiting Toxicities (DLTs) | 4 weeks
  Incidence and severity of dose-limiting toxicities (DLTs) following infusion of UCMYM802 injection at each dose level.

SECONDARY OUTCOMES:
Bio-distribution of UCMYM802 | 3 months
  CAR copies will be measured by qPCR to evaluate the expansion and persistence of CAR-T cells in vivo.
Peak Plasma Concentration (Cmax) | 3 months
  The maximum (peak) of CART cells observed in peripheral blood
Time to Maximum Plasma Concentration (Tmax) | 3 months
  The time for CART cells to reach maximum（peak）in peripheral blood
Area Under Curve (AUC) | 3 months
  The area under curve (AUC) from time zero to 24, 48 ,72 hours and AUC0-tlast, AUC0-inf in peripheral blood
Cytokine Level in Peripheral Blood | 2 years
  The concentration level of CAR-T cell related cytokines/chemokines in peripheral blood
Anti-drug Antibodies | 2 years
  Positive rate of anti-drug antibody in the serum of subjects
Objective Response Rate (ORR) | 2 years
  The proportion of subjects who achieved complete response (CR) or partial response (PR) according to the RECIST v1.1 criteria
Disease Control Rate (DCR) | 2 years
  The proportion of subjects who achieved complete response (CR), partial response (PR), or disease stability (SD) according to the RECIST v1.1 criteria
Duration of Response (DoR) | 2 years
  The time from the initial evaluation as complete remission (CR) or partial remission (PR) to the initial evaluation as disease progression (PD) or death from any cause
Progression-Free Survival (PFS) | 2 years
  The time from initial CART cell infusion to first disease progression (PD) or death for any cause
Overall Survival (OS) | 2 years
  The time from initial CART cell infusion to death due to any reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China